CLINICAL TRIAL: NCT04931641
Title: Improving Efficacy and Safety of Oral Iron Supplementation in HIV-infected Children by Providing Prebiotic Galacto-oligosaccharides As Adjunct Treatment: a Randomized Controlled Trial
Brief Title: Potential of Prebiotic Galacto-oligosaccharides in Improving Efficacy and Safety of Oral Iron Supplementation in HIV-infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fe-GOS-HIV
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Iron Deficiency; HIV
MeSH Terms: conditions — Iron Deficiencies | interventions — Prebiotics; maltodextrin; ferrous fumarate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 mg oral iron as ferrous fumarate (FeFum) with 7.5 g galacto-oligosaccharides (Experimental)
  Interventions: Dietary Supplement: Galacto-oligosaccharides; Dietary Supplement: Ferrous fumarate
- 50 mg oral iron as ferrous fumarate (FeFum) with 7.5 g maltodextrin (Placebo Comparator)
  Interventions: Other: Maltodextrin; Dietary Supplement: Ferrous fumarate

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharides — Prebiotic galacto-oligosaccharides (GOS)
  Other Names: Prebiotic
  Arms: 50 mg oral iron as ferrous fumarate (FeFum) with 7.5 g galacto-oligosaccharides
Other: Maltodextrin — Maltodextrin (placebo)
  Arms: 50 mg oral iron as ferrous fumarate (FeFum) with 7.5 g maltodextrin
Dietary Supplement: Ferrous fumarate — 50 mg iron as ferrous fumarate

SUMMARY:
The objectives of this randomized controlled trial in virally suppressed HIV-positive children with anemia and/or depleted iron stores are to determine the effect of prebiotic galacto-oligosaccharides (GOS) as adjunct treatment to 12 weeks of oral iron supplementation on:

1. iron status measured by conventional iron status biomarkers,
2. fractional absorption of iron (fraction of total body iron per day, measured as Kabs, the slope of 57Fe isotopic dilution) and mean total amount of iron absorbed each day (mg Fe/day, calculated as Kabs x mean total body iron),
3. systemic and gut inflammation, as well as gut mucosal integrity,
4. gut microbiome composition, and
5. adverse effects and gastrointestinal side-effects.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) in childhood can impair growth and cognition, as well as reduce school performance. Furthermore, anemia frequently complicates pediatric HIV infection and predicts disease progression and mortality. However, there is no international consensus on the treatment of ID and IDA in HIV-infected children, because of concerns around the efficacy and safety of oral iron supplements. Recent studies have suggested that oral iron supplements may increase gut inflammation in African children. This could be particularly detrimental in HIV-infected children, who may have gut immune activation, enteropathy and adverse shifts in the gut microbiome.

Previous stable iron isotope studies from the ETH Laboratory of Human Nutrition showed that the consumption of prebiotic galacto-oligosaccharides (GOS) together with supplemental doses of iron can increase iron absorption. In Kenyan infants, we further showed that the addition of GOS to an iron-containing micronutrient powder mitigated the adverse effects of iron on the gut microbiome.

Thus, we hypothesize that providing GOS as adjunct treatment to oral iron supplementation will improve efficacy (iron absorption and iron status), reduce systemic and gut inflammation, improve mucosal integrity, and mitigated iron-induced alterations in the gut microbiome, adverse events and gastrointestinal side-effects in virally suppressed HIV-infected children.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-15 years at baseline;
* Mild to moderate micro- and normocytic anaemia defined as Hb ≥8.0 and <11.5 / 12 g/dL (children 10-11 / 12-15 years) plus mean corpuscular volume ≤91.5 fL and/or iron deficiency defined as ferritin <30 µg/L or sTfR >8.3 mg/L;
* Body-Mass-Index-for-age Z-scores (BAZ) -3 to 2 SD of reference population;
* HIV criteria: HIV RNA viral load <50 copies/mL (measured as part of routine care);
* Willingness of caregiver to participate in the study;
* Caregiver speaks English, Afrikaans or isiXhosa;
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy) plus assent needs to be obtained from the child;
* Residence in the study area for the period of the study.

Exclusion Criteria:

* Child received iron supplements or antibiotic treatment 3 months prior to study start;
* Acute illness or other conditions that in the opinion of the PI or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol;
* Participants taking part in other studies involving medical or physical interventions.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Iron status: Serum Ferritin (ug/L) (SF) | 0, 6, 12 weeks
  Change in SF concentrations over the study period of 12 weeks
Iron status: Soluble Transferrin Receptor (mg/L) (sTfR) | 0, 6, 12 weeks
  Change in sTfR concentrations over the study period of 12 weeks
Iron status: Transferrin saturation (%) (Tsat) | 0, 6, 12 weeks
  Change in Tsat concentrations over the study period of 12 weeks
Iron status: Hemoglobin (g/dL) (Hb) | 0, 6, 12 weeks
  Change in Hb concentrations over the study period of 12 weeks
Fractional iron absorption | 0, 6, 12 weeks
  Fractional absorption of iron will be determined by measuring Kabs, the slope of 57Fe isotopic dilution over the study period. From this value, mean total amount of iron absorbed each day (mg Fe/day, calculated as Kabs x mean total body iron) can be estimated.

SECONDARY OUTCOMES:
Systemic inflammation: C-reactive protein (mg/L) (CRP) | 0, 6, 12 weeks
  Change in CRP concentrations over the study period of 12 weeks
Systemic inflammation: Alpha-1-acid glycoprotein (g/L) (AGP) | 0, 6, 12 weeks
  Change in AGP concentrations over the study period of 12 weeks
Hepcidin (nM) | 0, 6, 12 weeks
  Change in hepcidin concentrations over the study period of 12 weeks
Gut inflammation: Intestinal fatty acids binding protein (ng/ml) (IFABP) | 0 and 12 weeks
  Change in IFABP concentrations from baseline (0 weeks) to endpoint (12 weeks)
Gut inflammation: Fecal calprotectin (µg/g) | 0 and 12 weeks
  Change in fecal calprotectin concentrations from baseline (0 weeks) to endpoint (12 weeks)
Gut inflammation: Myeloperoxidase (µg /mL) (MPO) | 0 and 12 weeks
  Change in MPO concentrations from baseline (0 weeks) to endpoint (12 weeks)
Gut microbiome composition | 0 and 12 weeks
  Change in gut microbiome composition from baseline (0 weeks) to endpoint (12 weeks)
Fecal pH | 0 and 12 weeks
  Change in fecal pH from baseline (0 weeks) to endpoint (12 weeks)
HIV viral load (copies/ml) | 0 and 12 weeks
  Change in HIV viral load from baseline (0 weeks) to endpoint (12 weeks)
Gastrointestinal and respiratory symptoms | 12 weeks
  Self-reported gastrointestinal and respiratory symptoms assessed using a symptoms diary over the study period of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine Baumgartner, PhD, Principal Investigator — Swiss Federal Institute of Technology; Michael Zimmermann, MD, Study Chair — Swiss Federal Institute of Technology
Locations (1):
- Familiy Clinical Research Unit (FAMCRU), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No